CLINICAL TRIAL: NCT00042419
Title: Work and Health Disparities Among Rural Women
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 10939-CP-001
Record Dates: First submitted 2002-07-29; First posted 2002-08-01 (Estimated); Last update posted 2006-09-04 (Estimated); Status verified 2006-09

CONDITIONS: Tendonitis; Carpal Tunnel Syndrome; Cumulative Trauma Disorders; Overuse Syndrome
Keywords: Industrial Injuries; Tendonitis; Assembly Line
MeSH Terms: conditions — Tendinopathy; Carpal Tunnel Syndrome; Cumulative Trauma Disorders

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Prospective

SUMMARY:
This is a study of the effects of fast paced assembly line work on women. We are studying problems women in poultry processing have with their muscles, tendons, and nerves as well as acute injuries they have in the workplace. We are also studying how their work affects the quality of their lives.

ELIGIBILITY:
Women employed in poultry processing less than 9 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2002-03; Study Completion 2003-07

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States